CLINICAL TRIAL: NCT06351683
Title: Mito-LUTS: A Pilot Study of the Effect of MitoQ on Lower Urinary Tract Symptoms in Older Women With Metabolic Syndrome
Brief Title: Testing MitoQ on Lower Urinary Tract Symptoms in Older Women With Metabolic Syndrome
Acronym: Mito-LUTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Iman Al-Naggar, PhD (Other)
Collaborators: National Institute on Aging (NIA) (NIH); American Urological Association (Other); Urology Care Foundation (Unknown); Claude D. Pepper Older Americans Independence Center (OAIC) (Unknown)
Responsible Party: Sponsor-Investigator, Iman Al-Naggar, PhD, Assistant Professor, UConn Health
Organization: UConn Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-066-2; P30AG067988 (NIH)
Record Dates: First submitted 2024-04-01; First posted 2024-04-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Lower Urinary Tract Symptoms; Overactive Bladder Syndrome
Keywords: MitoQ; gerotherapeutics; urgency; urinary urgency; metabolic syndrome; aging; LUTS; OAB; geroscience
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Metabolic Syndrome | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded. Pharmacy will randomize and dispense capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MitoQ group (Experimental): 2x20mg MitoQ (mitoquinol mesylate) capsules taken orally daily before breakfast for 4 months
  Interventions: Drug: MitoQ (mitoquinol mesylate)
- Placebo Control group (Placebo Comparator): 2 placebo capsules taken orally daily before breakfast for 4 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MitoQ (mitoquinol mesylate) — MitoQ is an antioxidant molecule designed to target cell stress
  Other Names: MitoQ
  Arms: MitoQ group
Other: Placebo — Control capsules that contain all inactive ingredients found in the study drug capsules (i.e., placebo capsules do not contain mitoquinol mesylate)
  Arms: Placebo Control group

SUMMARY:
The goal of this clinical trial is to test the effect of a supplement called MitoQ (mitoquinol mesylate) on bladder symptoms such as urgency and frequency in women 50 years and older who have the metabolic syndrome. The main questions it aims to answer are:

* Is the study design feasible and acceptable to participants?
* Do participants taking the study drug get any improvement to their bladder symptoms compared to participants taking a placebo (a look-alike substance that contains no drug)?

Participants will take 2 capsules of the study drug every morning for 4 months, answer many questions about their health including questions about their bladder health, perform physical and cognitive testing, give blood and urine samples, collect urine over 24 hour periods 3 times over the 4 months of the study, complete 3 day bladder diaries about how much they drink and void, undergo electrocardiograms, have their vitals and measurements (weight, height, waist circumference) taken, participate in 4 visits to the clinical research area and participate in many phone calls of varying length. Researchers will compare participants who were taking capsules containing MitoQ and participants taking capsules not containing MitoQ to see if MitoQ improves their bladder symptoms (urgency, frequency, nocturia, incontinence, etc.)

DETAILED DESCRIPTION:
Both aging and the metabolic syndrome are risk factors for lower urinary tract symptoms (LUTS, including urgency, frequency, nocturia (nighttime urination), and incontinence). This study aims to test whether an oral supplement that targets biological aging pathways can improve lower urinary tract symptoms (LUTS) in women aged 50 years and older with the metabolic syndrome (a cluster of conditions that occur together, increasing the risk of heart disease, stroke and type 2 diabetes). MitoQ, a strong mitochondrial-targeted antioxidant molecule, has been shown to target mitochondrial dysfunction, oxidative stress, inflammation, and endothelial dysfunction, all aging pathways that are also found to be dysregulated in conditions that cause LUTS such as the overactive bladder syndrome. Women aged 50 years and older who have the metabolic syndrome per the new International Diabetes Federation (IDF) definition and have had urinary urgency for at least 3 months will be invited to participate in the study. They will be screened by phone for major study inclusion/exclusion criteria and then invited for an in-person screening visit where blood will be drawn and measurements taken to confirm eligibility. Once eligible, participants will be randomly assigned to MitoQ or placebo (2MitoQ:1placebo) and asked to take 2 capsules daily (40mg MitoQ total) 30 minutes before breakfast for 4 months. Participants will come back for study visits at 8 and 16 weeks, and will receive two study data collection phone calls at 4 and 12 weeks, where they will answer questions about their bladder. There will be many other shorter phone calls throughout the study to check for adherence and adverse events. In addition to questionnaires assessing bladder function, participants will undergo tests of frailty, physical function, cognitive function and asked many questions about their health and medication. We will also draw blood for safety assessment and to measure aging molecules in the blood at each visit and see whether they change with treatment. Urine will also be collected at each study visit and participants will be asked to collect urine at home (first morning and 24-hour urine) and bring it to each of their study visits, which will be used for measuring aging molecules and testing how they change with the study drug. Participants will also fill out three-day voiding diaries to provide information about their voiding and LUTS.

ELIGIBILITY:
Inclusion Criteria

The new IDF's 2006 consensus worldwide definition for MetS will be followed for inclusion. MetS will be defined as having central obesity with ethnicity-specific values, plus two or more of the following criteria: Hypertension, dyslipidemia, or hyperglycemia. Hypertension is defined by the use of antihypertensive medication and/or blood pressure of ≥130/85 mmHg. Dyslipidemia is defined as blood triglycerides >150mg/dL or high-density lipoprotein (HDL) < 50mg/dL, or specific treatment for either lipid abnormality. Hyperglycemia is defined as a fasting glucose ≥100mg/dL. Inclusion criteria for LUTS are having urgency with or without other urinary symptoms for at least 3 months, with a score of 1 or 2 on the Urgency Perception Scale questionnaire 60 , and a total score of at least 6 on the OABSS questionnaire (with at least a score of 2 on the third OABSS question "How often do you have a sudden desire to urinate, which is difficult to defer?").

* Women 50years or older with metabolic syndrome and LUTS as defined above.
* Speak, read and understand English
* Willingness to provide consent and participate in all aspects of the trial including randomization to the intervention group

Exclusion Criteria

The exclusion criteria for Mito-LUTS include conditions that will interfere with our research questions, including advanced co-morbidities and immunological disorders. They are as follows:

* Frailty, defined as meeting 3 of 5 frailty indicators of the Fried Frailty Phenotype
* History of severe renal impairment and/or eGFR ≤ 60 mL/min/1.73m2 at the study physician's discretion
* Excessive alcohol use (more than 14 alcoholic drinks/week)
* Clinical/laboratory evidence of hepatic disease (via medical history and/or AST and/or ALT ≥ 3 times upper limit of normal at screening)
* Poorly Controlled Diabetes
* Unwilling or unable (due to significant cognitive impairment) to provide informed consent.
* Terminal illness with life expectancy less than 12 months
* Advanced neurological disorder (Alzheimer's, Parkinson's, ALS, MS, dementia, seizures)
* A score of 30 or less on the modified Telephone Screening of Cognitive Status administered during the in-person screening visit.
* Cancer or history of gynecological cancer or history of cancer requiring chemotherapy or radiation.
* A history of gastric ulcers.
* Abnormal findings on endoscopy.
* Recent (within the last 2 weeks) or current chronic use of NSAIDs or other drugs or agents with the potential for gastric mucosal toxicity (except for daily use of baby aspirin or famotidine for which participants will not be excluded). Sporadic use of NSAIDs will not be an exclusion criterion.
* Significant co-morbid disease (severe chronic obstructive pulmonary disease, active rheumatologic diseases, chronic infection (HIV, tuberculosis), severe congestive heart failure (NYHA class 4), myocarditis, etc)
* Myocardial infarction, stroke or hospitalization for heart failure in the last 12 months
* QTc >460 ms at screening on ECG
* Prior diagnosis of ventricular arrhythmia (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
* Severe active psychiatric disorder (e.g. bipolar, schizophrenia)
* Unable to complete physical performance testing due to medical conditions (at discretion of the PI)
* Unintentional weight loss >15 lbs in past 12 months
* Immunosuppressive disorders or taking immunosuppressive medications (including oral prednisone > 10mg/day)
* Sub-cerebellar lesions
* Subjects must not be on warfarin or other blood thinning medications or have a known bleeding disorder.
* Conditions that might interfere with clinical diagnosis (such as pelvic organ prolapse ≥ stage 2, pelvic radiotherapy, any concurrent condition that could cause incontinence, hematuria, vaginitis, neurogenic lower urinary tract dysfunction); chronic pelvic pain syndrome, interstitial cystitis/bladder pain syndrome, pelvic malignancy, active urinary tract infection (UTI), recent urologic procedure (<6 months).
* Clean intermittent catheterization or indwelling catheter
* Current participation in another interventional study
* Pregnancy and nursing
* Subjects must not have used antibiotics for at least 3 weeks prior to visit 1, received a vaccination in the 2 weeks prior to visit 1 or used medicine that alters the immune response (eg high dose corticosteroids) in the 6 months prior to visit 1. Subjects must not have had an acute infection in the 3 weeks prior to visit 1 or had a major severe illness or been hospitalized in the 3 months prior to visit 1. If participants are within any of these windows when they are screened, they will be scheduled for a screening visit but will only be invited for Visit 1 after these specified windows have elapsed and/or infections have resolved.
* Subjects must not be on or have taken any of the following anti-muscarinics or β3- adrenoreceptor agonists for 3 weeks prior to visit 1: o Darifenacin (enablex), Oxybutynin (ditropan), Solifenacin (vesicare), Fesoterodine (Toviaz), Tolterodine (detrol), Trospium (sanctura), Imipramine (tofranil), Mirabegron (myrbetriq), Vibegron (gemtesa)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sex assigned at birth is Female
Enrollment: 50 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder Symptom Score (OABSS) | Week 0, Week 4, Week 8, Week 12, Week 16
  The OBSS is a validated bladder symptom questionnaire routinely used in assessing lower urinary tract symptoms and overactive bladder syndrome.
  The OABSS questionnaire consists of 4 questions and has a minimum score of 0 and a maximum score of 15.
  Scores on the OABSS of ≤5 are defined as mild, those of 6-11 as moderate, and those of ≥12 as severe LUTS.

SECONDARY OUTCOMES:
Three-day bladder voiding diary | Week 0, Week 8, Week 16
  Participants will record times and amounts of liquids ingested and urine produced for 3 days. They will also record their urge at each voiding instance and incontinence episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Iman M Al-Naggar, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States